## Kinesiotaping in Lateral Epicondylitis (NCT03074500)

(Unique Protocol ID: 09.2017.004)

## STATISTICAL PLAN

IBM SPSS Statistics for Windows, Version 20,0 (Armonk, NY, USA) will be used to perform all of the analysis. Statistical significance is accepted as p<0.05. The histogram and normality plots and Shapiro-Wilk normality test will be used to evaluate the distribution of variables prior to test selection. Descriptive statistics will be presented as median (25–75%) for the nonnormally distributed quantitative and ordinal data and number (minimum-maximum) for the categorical variables. Friedman test will be used to establish within group changes over time in outcome variables. Wilcoxon's signed-rank test will be performed to show differences in the parameters between baseline and follow-up points. Between groups differences will be analyzed by using Kruskal Wallis test. Results will be considered significant when p < 0.05. The Mann-Whitney U test will be used to analyze the significance of pairwise differences using the Bonferroni correction (post-hoc test) to adjust for multiple comparisons when an overall significance significance is observed. Using the Bonferroni correction, a p value of less than 0.017 (0.05/3) will be considered statistically significant. Effect sizes (ES) wil be calculated by using GPower V.3.1.7 (University of Kiel, Kiel, Germany) as previously described by Guo et al. The effect sizes will generally be defined as small (r=0.1), median (r= 0.3), and large (r=0.5) (Fritz CO, 2012).